CLINICAL TRIAL: NCT06210607
Title: A Phase I, Randomized, Double-Blind, Placebo-Controlled Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of Single and Multiple Doses of HS-10511 in Healthy Subjects
Brief Title: A Trial of HS-10511 in Healthy Subjects
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Jiangsu Hansoh Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HS-10511-101
Record Dates: First submitted 2024-01-08; First posted 2024-01-18 (Actual); Last update posted 2024-01-18 (Actual); Status verified 2024-01

CONDITIONS: Hypertrophic Cardiomyopathy
Keywords: Cardiomyopathy; Hypertrophy; Heart Diseases; Cardiovascular Diseases
MeSH Terms: conditions — Cardiomyopathy, Hypertrophic; Cardiomyopathies; Hypertrophy; Heart Diseases; Cardiovascular Diseases

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HS-10511 Tablets (Experimental): Subjects will be assigned to one of 5~6 planned dose cohorts in (single ascending dose)SAD and one of 4 planned dose cohorts in (multiple ascending dose)MAD.
  Interventions: Drug: HS-10511 Tablets
- HS-10511 Tablets Placebo (Placebo Comparator): Subjects will be assigned to one of 5~6 planned dose cohorts in SAD and one of 4 planned dose cohorts in MAD.
  Interventions: Drug: HS-10511 Tablets Placebo

INTERVENTIONS:
Drug: HS-10511 Tablets — HS-10511 tablets for 5~6 SAD cohorts and 4 MAD cohorts
  Arms: HS-10511 Tablets
Drug: HS-10511 Tablets Placebo — HS-10511 tablets placebo for 5~6 SAD cohorts and 4 MAD cohorts
  Arms: HS-10511 Tablets Placebo

SUMMARY:
This study is a phase I, randomized, double-blind, placebo-controlled clinical trial evaluating the safety, tolerability, and pharmacodynamic (PK) and pharmacodynamic (PD) characteristics of HS-10511 when administered as single oral dose and multiple oral doses in healthy adult subjects.

DETAILED DESCRIPTION:
This study is a phase I, randomized, double-blind, placebo-controlled clinical trial evaluating the safety, tolerability, and PK and PD characteristics of HS-10511 in healthy adult subjects. This study consists of two parts: Part 1 is a single ascending dose (SAD) peroid in healthy subjects and Part 2 is a multiple ascending dose (MAD) period. Each period is composed of the screening, baseline, dosing and observation, and follow-up periods. All subjects will sign a written informed consent form (ICF) and will be assessed for eligibility criteria before entering the screening period (D-28-D-1). Subjects who meet all inclusion criteria and none of the exclusion criteria will be admitted in the baseline period (i.e., 1 day before dosing, D-1), undergo baseline assessment and randomization, complete dosing and the safety, tolerability, and PK and PD assessments within the given time period, and complete outpatient visits at the given follow-up time after discharge.

ELIGIBILITY:
Inclusion Criteria:

* Healthy males or females aged 18-45 years (inclusive) at screening;
* Body weight ≥ 50 kg in males and ≥ 45 kg in females, and body mass index (BMI): 18.0-27.9 kg/m2 (inclusive) at screening;
* Acoustic windows are adequate for performing precise transthoracic echocardiography;
* Normal cardiac structure and function as determined by a cardiologist, or presence of clinically irrelevant abnormalities at the discretion of a cardiologist or ultrasound specialists;
* Normal clinical laboratory test results at screening and admission to the clinical study site, or presence of clinically irrelevant abnormalities at the discretion of the investigator;
* Able to understand and agree to sign the ICF, and to agree to follow all study procedures and restrictions (including remaining at the study site within the time period defined in the schedule of assessments);
* Willing to and able to perform normal non-vigorous physical activities starting from 48 h before D-1, during the admission to the study site, and even during the study period;
* Able to sufficiently understand the study content, process, and potential adverse reactions, and voluntarily sign the ICF.

Exclusion Criteria:

* Those with possibly clinically relevant diseases are not suitable for participating in this study as assessed by the investigator at screening;
* Previous history of syncope, history of clinically significant cardiac disease including;
* Presence of a medical history of malignancy of any type within 5 years before screening;
* Consumption of caffeine-and/or xanthine-rich food or beverages (e.g., coffee, tea, chocolate, and caffeine-containing carbonated beverages such as cola), tobacco-containing products (e.g., cigarettes), and alcohol or alcoholic products within 48 h before dosing;
* Consumption of grapefruit, grapefruit juice, seville orange, seville orange jam, and seville orange juice or other grapefruit- or seville orange-containing products within 7 days before the first dose;
* Positive breath alcohol test or presence of a history of heavy smoking or alcoholism within 6 months before screening: heavy smoking (more than 5 cigarettes or the equivalent amount of tobacco per day); alcoholism (≥ 14 units of alcohol per week: 1 unit = 285 mL of beer, 25 mL of spirits with an alcohol by volume of ≥ 40%, or 150 mL of wine);
* Positive urine drug test or abuse of barbiturates, amphetamines, benzodiazepines, cocaine, opiates, marijuana, methadone, phencyclidine, and tricyclic antidepressants or methamphetamines, or other situation that is unfit to participate in the study judged by the researcher;
* Subject has a positive serum β-human chorionic gonadotropin (β-hCG) test at screening, or is in pregnancy, or is in lactation;
* Presence of clinically relevant gastrointestinal complaints, a history of gastrointestinal diseases (e.g., Crohn's disease, and ulcerative colitis), or a history of surgeriesthat may affect the absorption of the investigational drug within 7 days before the first dose;
* Those with a history of any serious drug hypersensitivity, allergic diseases (e.g., asthma, severe urticaria, and severe allergic rhinitis), or other allergic constitutions are not suitable for participating in this study at the discretion of the investigator;
* Other conditions or causes that make subjects unsuitable for participating in this clinical study, as determined by the investigator.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — No less than 1/3 of either gender
Enrollment: 96 (Estimated)
Dates: Start 2024-01-31 (Estimated); Primary Completion 2024-06-30 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
The incidence and severity of adverse events (AE), serious adverse events (SAE) and adverse events leading to withdrawal from the trial and the correlation with the investigational drug in single ascending dose (SAD) | Day 1 to day 8
  The definition of adverse event [AE] is any untoward medical occurrence in a patient or clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. The definition of serious adverse event [SAE] is any untoward medical occurrence at any dose that results in death; is life threatening; requires inpatient hospitalization or prolongation of existing hospitalization; results in persistent disability/incapacity; results in congenital anomaly/birth defect.
Number of participants with clinically significant change from baseline in vital signs in SAD | Day 1 to day 8
Number of participants with clinically significant change from baseline in 12-lead electrocardiogram (ECG) findings in SAD | Day 1 to day 8
Number of participants with clinically significant abnormalities in laboratory examination in SAD | Day 1 to day 8
Number of participants with clinically significant abnormalities in physical examination in SAD | Day 1 to day 8
The incidence and severity of adverse events (AE), serious adverse events (SAE) and adverse events leading to withdrawal from the trial and the correlation with the investigational drug in multiple ascending dose (MAD) | Day 1 to Day 14
  The definition of adverse event [AE] is any untoward medical occurrence in a patient or clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. The definition of serious adverse event [SAE] is any untoward medical occurrence at any dose that results in death; is life threatening; requires inpatient hospitalization or prolongation of existing hospitalization; results in persistent disability/incapacity; results in congenital anomaly/birth defect.
Number of participants with clinically significant change from baseline in vital signs in MAD | Day 1 to Day 14
Number of participants with clinically significant change from baseline in 12-lead electrocardiogram (ECG) findings in MAD | Day 1 to Day 14
Number of participants with clinically significant abnormalities in laboratory examination in MAD | Day 1 to Day 14
Number of participants with clinically significant abnormalities in physical examination in MAD | Day 1 to Day 14